CLINICAL TRIAL: NCT06237712
Title: Explorative Study to Investigate the Acid-base Response to Sodium and Potassium Salts in Patients With Chronic Kidney Disease.
Acronym: 5S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ewout Hoorn, Prof. dr. Ewout Hoorn, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL84462.078.23
Record Dates: First submitted 2023-07-25; First posted 2024-02-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Metabolic Acidosis; CKD; Electrolyte and Fluid Balance Conditions
MeSH Terms: conditions — Acidosis

STUDY DESIGN:
Intervention Model Description: Single-center, placebo-controlled double-blind randomized crossover study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Sodium chloride (Active Comparator): 40 mmol of oral sodium chloride daily for 5 days
  Interventions: Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of sodium chloride
- Sodium bicarbonate (Active Comparator): 40 mmol of oral sodium bicarbonate daily for 5 days
  Interventions: Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of sodium bicarbonate
- Potassium chloride (Active Comparator): 40 mmol of oral potassium chloride daily for 5 days
  Interventions: Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium chloride
- Potassium bicarbonate (Active Comparator): 40 mmol of oral potassium bicarbonate daily for 5 days
  Interventions: Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium bicarbonate
- Potassium gluconate (Active Comparator): 40 mmol of oral potassium gluconate daily for 5 days
  Interventions: Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium gluconate
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo caps

INTERVENTIONS:
Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium chloride — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Potassium chloride
Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium gluconate — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Potassium gluconate
Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of potassium bicarbonate — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Potassium bicarbonate
Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of sodium chloride — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Sodium chloride
Dietary Supplement: Dietary supplement consisting of 40 mmol/daily of sodium bicarbonate — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Sodium bicarbonate
Dietary Supplement: Placebo caps — The supplements are delivered in plain vegetable 00 caps, stabelizing additives are potatostarch, sunflower lecithine and sunflower oil. The capsuels are free of titanium oxide and suited for human consumption.
  Arms: Placebo

SUMMARY:
With this research the investigators want to study how patients with chronic kidney disease respond to different sodium- and potassium salts. Potassium salts can prevent kidney damage and cardiovascular disease, however patients with chronic kidney disease can responds differently. Extra potassium can increase the amount of potassium in the blood and extra chloride can cause acidosis. With this study the investigators will gain more insight in how patients with chronic kidney disease respond to sodium and potassium salts and which one is more favorable.This information can then be used to guide the application of salt substitutes and dietary adjustments in patients with chronic kidney disease.

DETAILED DESCRIPTION:
Rationale: Patients with chronic kidney disease (CKD) consume a low potassium diet which is associated with progressive CKD and cardiovascular disease. Increasing dietary potassium intake to recommended levels may therefore improve cardiorenal outcomes, but the response to increased potassium intake in patients with CKD is unclear. Therefore, the investigators recently tested the response to 40 mmol potassium chloride in patients with CKD and showed that this is generally well-tolerated. However, patients did develop mild hyperchloremic metabolic acidosis, which may offset the beneficial effects of potassium. The investigators hypothesize that this is a form of chloride-induced acidosis that may be prevented by giving potassium with a different anion than chloride. To further investigate this, the investigators propose to test the response to five different sodium and potassium salts in patients with CKD. These results should inform us on how to best correct a potassium-deficient diet in patients with CKD.

Objective: To test the effects of five different sodium and potassium salts in patients with CKD.

Study design: Investigator-initiated, single-center, placebo-controlled double-blind randomized crossover study.

Study population: Adult outpatients (age ≥ 18 years) with CKD stage G3b or G4 using renin-angiotensin-aldosterone system inhibitors (RAAS-I).

Intervention: Capsules with 40 mmol potassium chloride, potassium bicarbonate, potassium gluconate, sodium bicarbonate, sodium chloride or placebo (3 x 3 capsules per day).

Main study parameters/endpoints: Difference in plasma bicarbonate after treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The study lasts 6 weeks and consists of 7 visits that will consist of blood sampling, 24-hour urine collection and spot urine collection. We will also provide an automated blood pressure measuring device for at home blood pressure measurements. Although these procedures are time-consuming and may be experienced as burdensome, they are all routine clinical measurements and safe. Patients may experience a pill-burden. The two risks of the salt supplements are hyperkalemia (with potassium salts) and hypertension (with sodium salts). Based on our previous studies a minority of patients is expected to develop these side-effects (< 12%). Safety measures to prevent, monitor and treat these side-effects are included in the study protocol. There are no direct benefits for patients participating in this trial, but the results will contribute to a better understanding on the feasibility of dietary modifications and salt substitution in patients with CKD to improve health. Patients will be reimbursed for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* CKD G3b or G4 (44 - 15 ml/min/1.73 m2)
* Use of RAAS-I (ACE-inhibitor or angiotensin receptor blocker, ARB)

Exclusion Criteria:

* Use of any of the following drugs or supplements: mineralocorticoid receptor antagonists, potassium-sparing diuretics, oral potassium binders, immunosuppressive medication, tolvaptan, acetazolamide, topiramate, sodium bicarbonate.
* Patients using double RAAS blockade (i.e., ACE-inhibitor + ARB).
* Metabolic alkalosis (plasma bicarbonate >27 mmol/L) at last outpatient visit
* Kidney transplant recipients
* Patients with an active gastro-intestinal ulcer
* Patients with previous history of ventricular cardiac arrhythmia
* Patients with a life expectancy < 6 months
* Incapacitated subjects or subjects who are deemed unfit to adequately adhere to instructions from the research team
* Women who are pregnant, breastfeeding or consider pregnancy in the coming 7 weeks
* Patients with chronic respiratory acidosis in previous medical history
* Hyperkalemia (plasma potassium >5.5 mmol/L) at V0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Plasma bicarbonate by blood draw | After 5 days of intervention
  The absolute difference per treatment group in measured plasma bicarbonate after treatment.
  After each treatment of 5 days, plasma bicarbonate will be measured by blood sampling.
  The difference between the groups (treatments) will be the main outcome and comparator.

SECONDARY OUTCOMES:
Plasma electrolyte levels | After 5 days of intervention
  Na, Cl, K, Mg, Ca, Phosphate (all in mmol/L)
Urinary citrate | After 5 days of intervention
  Urinary citrate in mmol/24h
Urinary ammonia | After 5 days of intervention
  urinary ammonia in mmol/24, calculated using the Berthelot method
Titratable acid | After 5 days of intervention
  Titratable acid = (0.067) × (mLs NaOH (sample titration) - mLs NaOH (blank titration)) × 75/ mLs of sample
Net acid excretion | After 5 days of intervention
  Net acid excretion unit/24h, formula = sum of the titratable acid and concentration of ammonia minus the concentration of bicarbonate.
Potential renal acid load | After 5 days of intervention
  PRAL (mEq/d) = 0.49 × protein (g/d) + 0.037 × phosphate (mg/d) - 0.021 × potassium (mg/d) - 0.026 × magnesium (mg/d) - 0.013 × calcium (mg/d).
Body weight | After 5 days of intervention
  Weight measured by a scale in kilograms
Blood pressure | 2 measurements in the morning and evening for 5 days per treatment repeated for 6 treatments in total
  Systolic and diastolic blood pressure measured 2 times daily during the study, so 20 times during the 5 days of supplement usage. Measurements will be done in the morning and evening measured twice in seated position with an automatic blood pressure monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No